CLINICAL TRIAL: NCT04905446
Title: Measurement of NAD+ Synthesis in Human Skeletal Muscle
Acronym: NAD-flux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1581811
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Skeletal Muscle
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy male subjects (Other)
  Interventions: Other: Deuterated nicotinamide (D4-NAM) IV infusion; Procedure: Skeletal muscle biopsy; Procedure: Skin tissue biopsy

INTERVENTIONS:
Other: Deuterated nicotinamide (D4-NAM) IV infusion — Nicotinamide adenine dinucleotide (NAD) is a vitally important substance that is found in all cells of the body. D4-NAM (in normal saline) will be infused via an indwelling catheter.The IV infusion will continue for 8 hrs.
Procedure: Skeletal muscle biopsy — Participants will have a muscle biopsy performed on the muscle in the thigh. We will collect a small sample of blood before the biopsy. This procedure is used to sample muscle cells from the right or left leg Vastus Lateralis (thigh) muscle.
Procedure: Skin tissue biopsy — This procedure is used to sample skin tissue from the upper thigh via a punch biopsy.

SUMMARY:
The key objective of this pilot research study is to dose human volunteers with a heavy (non-radioactive) isotope derivative of nicotinamide to detect NAD synthesis in human skeletal muscle. The ultimate goal is to examine the impact of lifestyle choices, aging, nutraceuticals, and drugs on the rate of NAD synthesis in human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects who, at the time of screening are between the ages of 21 to 40 years of age, inclusive.
2. BMI between 20-30 kg/m2 at the screening visit (SV)
3. Understands the procedures and agrees to participate by giving written informed consent
4. Willing and able to comply with the scheduled study day and other study procedures

Exclusion Criteria:

Acute or chronic medical conditions or medication that would contraindicate the participation in the research testing or could potentially affect metabolic function including, but not limited to:

1. History of type 1 or type 2 diabetes mellitus, including pre-diabetes (HbA1c > 5.7)
2. History of any antihyperglycemic agent (e.g., insulin)
3. Currently taking medications that can alter glucose homeostasis (e.g., steroids, glucocorticoids, nicotinic acid) or skeletal muscle metabolism
4. History of taking Tru Niagen, Basis (or any other NR-containing NAD+ booster) or niacin supplements.
5. Any bleeding disorders
6. Currently taking any aspirin (ASA) (including baby ASA) or NSAIDs (ibuprofen, naproxen, etc.) that cannot be safely stopped throughout the study. There is a recommended hold on NSAIDs and/or ASA for at least 2 days prior to biopsy, although not exclusionary
7. Presence of bruising in lower extremities
8. Any major surgery within the past 3 months
9. Any acute or chronic infections
10. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological or allergic diseases, but excluding untreated, asymptomatic, seasonal allergies at the time of intervention.
11. Previous difficulty with lidocaine or other local anesthetic agents
12. Thyroid dysfunction (suppressed TSH, elevated TSH <10 µIU/ml if symptomatic or elevated TSH >10 µIU/ml if asymptomatic)
13. Uncontrolled hypertension (BP >160 mmHg systolic or >100 mmHg diastolic)
14. Use of tobacco or nicotine-containing products within the last 12 months.
15. Chronic kidney disease with GFR of < 60
16. Anemia (hemoglobin <12 g/dl) during screening
17. History of human immunodeficiency virus (HIV), hepatitis B or hepatitis C
18. Liver function testing for ALT or AST greater than or equal to 2 times the upper limit of normal
19. Participation in studies involving investigational drug(s) within 30 days prior to Screening visit
20. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to Screening (participants may not donate blood any time during the study, through the final study day)
21. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study days Labs may be repeated at the discretion of the PI, MI or Sub-investigators (Sub-I).

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Measurement of NAD+ mass isotopomers in extracts from human muscle and skin tissue biopsies as determined by liquid chromatography-mass spectrometry (LC-MS) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gardell, PhD, Principal Investigator — Senior Investigator, Translational Research Institute, AdventHealth
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States